CLINICAL TRIAL: NCT05426200
Title: Pre-transplant Health Coaching to Improve Patient-Reported Outcomes in Lung Transplant Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-002675
Record Dates: First submitted 2022-05-05; First posted 2022-06-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lung Transplant
Keywords: Self-management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): Patient will work with a health coach to improve self-management skills, and receive usual pre-transplant education.
  Interventions: Behavioral: Health Coaching
- Control (No Intervention): Patients will receive usual pre-transplant education.

INTERVENTIONS:
Behavioral: Health Coaching — Patients will work with a health coach by telephone for up to 12 sessions over a 12-16 week period.
  Arms: Health Coaching

SUMMARY:
To examine the effectiveness of an individual health coaching intervention for lung transplant candidates. This intervention will include up to 12 health coaching sessions via phone call over a 12-16 week period. This will be compared to a usual care group the receives pre-transplant care and education alone.

ELIGIBILITY:
Inclusion Criteria:

* Waitlisted or deferred for lung transplantation at Mayo Clinic Rochester, Mayo Clinic Florida, or University of Washington

Exclusion Criteria:

* Under 18 years old
* Non-English speaking, nonverbal, or extremely hard of hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Score on Chronic Respiratory Disease Questionnaire (CRQ) Mastery Subdomain | Baseline, 12-16 Week Follow-up
  Participants will complete questions comprising the CRQ Mastery subdomain (7,10,13, and 19) of a 20-item Chronic Respiratory Questionnaire (CRQ) at baseline and after the 12-week intervention. CRQ Mastery subscores measure self-management abilities and range from 1 to 7, with higher scores indicating higher self-efficacy. The minimum clinically important difference is 0.5.
Change in Score on Chronic Respiratory Disease Questionnaire (CRQ) Emotional Function Subdomain | Baseline, 12-16 Week Follow-up
  Participants will complete questions comprising the CRQ Emotional Function subdomain (6,9,12,14,16,18, and 20) of a 20-item Chronic Respiratory Questionnaire (CRQ) at baseline and after the 12-week intervention (or 12-16 weeks from baseline). CRQ Emotional Function subscores measure emotional health and range from 1 to 7, with higher scores indicating better emotional health. The minimum clinically important difference is 0.5.

SECONDARY OUTCOMES:
Post-Transplant Quality of Life Chronic Respiratory Disease Questionnaire (CRQ) Composite | Post-Transplant Follow-up, on Average 1 Year
  Participants will complete a 20-item Chronic Respiratory Questionnaire (CRQ) at baseline and at three to six months post-transplant. CRQ composite scores measure health-related quality of life and range from 4 to 28, with higher scores indicating better QOL. The minimum clinically important difference is 2.0. The intervention (or control) phase is 12-16 weeks, but patients will be followed until they are one-year post-lung transplant. Since timing of lung transplant is unknown, the timing of this measurement could range from months to several years after enrollment.
Intervention Feasibility and Acceptability via Qualitative Surveys and Interviews | 12-16 Week Follow-up
  Acceptability and feasibility of the intervention will be examined via qualitative surveys (Likert scale rated questions and open-ended questions) and, for a subset of participants, semi-structured qualitative interviews. This qualitative data will assess the timing, duration, and number of health coaching sessions; any technical issues; the degree of therapeutic alliance with the assigned health coach; the participants' opinions of the perceived benefits of the intervention; and participant input regarding any needed changes in the design for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Cassie C Kennedy, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No